CLINICAL TRIAL: NCT02411513
Title: Open-trial on the Acute Treatment of Migraine Using the CEFALY Device
Brief Title: Acute Treatment of Migraine Using the CEFALY Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50208
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): 60 minutes of CEFALY stimulation as acute treatment of an on-going attack
  Interventions: Device: CEFALY

INTERVENTIONS:
Device: CEFALY

SUMMARY:
The purpose of this study is to investigate the efficacy of e-TNS with the Cefaly® device as an acute treatment for a migraine attack. This open clinical trial will study the acute treatment of migraine using the Cefaly® device, prior to development of a sham-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a history of episodic or chronic migraine with or without aura, meeting the diagnostic criteria listed in ICHD-III beta (2013) section 1, migraine (1), with the exception of ''complicated migraine'' (i.e., hemiplegic migraine, migraine with brainstem aura, ophthalmoplegic migraine- recurrent painful ophthalmoplegic neuropathy, migrainous infarction)
* The patient must be experiencing a migraine attack lasting for at least 3 hours, with pain intensity stabilized for at least 1 hour. The location of the headache should be frontal, retro- or peri- orbital, on one or either side.

Exclusion Criteria:

* Pregnant women
* Patients having received treatment with onabotulinum toxin (e.g., Botox, Dysport, Xeomin) to the head in the prior 4 months
* Patients having received supraorbital nerve blocks in the prior 4 months
* Diagnosis of other primary or secondary headache disorders, except of Medication Overuse Headache
* Patients with only temporal or occipital headaches
* Patients taking opioid medications
* Patients having taken abortive migraine medication in the prior 3 hours
* Allodynia: intolerance to supraorbital neurostimulation (allodynia) that makes the treatment not applicable (the patients will be excluded while the neurostimulation has already started).
* Implanted metal or electrical devices in the head
* Cardiac pacemaker or implanted or wearable defibrillator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change of pain intensity at 1 hour (VAS score) | 1 hour
  Mean change in intensity of pain at 1 hour when compared to baseline, measured on a visual analog scale (VAS) ranging from 0 to 11

SECONDARY OUTCOMES:
Change of pain intensity at 2 hours (VAS score) | 2 hours
  Mean change in intensity of pain at 2 hours when compared to baseline, measured on a visual analog scale (VAS) ranging from 0 to 11
Patients with no need of medication at 2 hours | 2 hours
  Percentage of patients not having required rescue medication after 2 hours
Patients with no need of medication at 24 hours | 24 hours
  Percentage of patients not having required rescue medication after 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Headache Center, New York, New York, United States